CLINICAL TRIAL: NCT05107908
Title: Neuronal and Behavioral Effects of an Implicit Priming Approach to Improve Eating Behaviors in Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20-2821; R01DK125417 (NIH)
Record Dates: First submitted 2021-11-03; First posted 2021-11-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Overweight and Obesity
Keywords: Eating; Overweight; Obesity; Food; Weight Loss; Magnetic Resonance Imaging; Neuroimaging; Brain; Body Weight
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Implicit Priming (Experimental): Participants will complete active implicit priming, in which food images are implicitly primed (i.e., below conscious awareness) with images of positive or negative affect. This will be completed on a weekly basis for 12 weeks, for approximately 10 minutes each time.
  Interventions: Behavioral: Active Implicit Priming
- Control Implicit Priming (Placebo Comparator): Participants will complete control implicit priming, which matches the active intervention, but with neutral stimuli as primes. This will be completed on a weekly basis for 12 weeks, for approximately 10 minutes each time.
  Interventions: Behavioral: Control Implicit Priming
- Food Exposure Task (Active Comparator): Participants will complete a Food Exposure Task, in which they will be asked to smell, feel, lick, and imagine eating food items, but without actually eating them. This will be completed on a weekly basis for 12 weeks, for approximately 10-30 minutes each time.
  Interventions: Behavioral: Food Exposure Task

INTERVENTIONS:
Behavioral: Active Implicit Priming — Approximately 10-minute behavioral intervention
  Arms: Active Implicit Priming
Behavioral: Control Implicit Priming — Approximately 10-minute behavioral intervention
  Arms: Control Implicit Priming
Behavioral: Food Exposure Task — Approximately 10-30 minute behavioral intervention
  Arms: Food Exposure Task

SUMMARY:
The purpose of this study is to determine how different behavioral interventions designed to alter food perceptions and behaviors affect brain responses to food, eating behaviors, and body weight.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* BMI of 27 or greater

Exclusion Criteria:

* MRI contraindications (e.g., metal or electronic devices in the body)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Blood Oxygen Level Dependent (BOLD) Response to Visual Food Cues as Measured by Functional Magnetic Resonance Imaging | Baseline, 12 weeks
  Percent change in blood oxygen level dependent (BOLD) response from baseline to after the 12-week intervention while viewing visual food cues will be measured using functional magnetic resonance imaging (fMRI), focusing on insula, striatum, and prefrontal cortex.
Change in Food Image Ratings | Baseline, 12 weeks
  Food image ratings change from baseline to after the 12-week intervention. Food images are rated on "desire to eat" by visual analogue scale (0-100), with higher scores indicating greater desire to eat.
Change in Food Intake | Baseline, 12 weeks
  Food intake change from baseline to after the 12-week intervention. Food intake will be measured as total calories consumed during an ad libitum meal.

SECONDARY OUTCOMES:
Percent Change in Body Weight | Baseline, 12 weeks
  Percent change in body weight (kg) from baseline to after the 12-week intervention.
Change in Fat Mass | Baseline, 12 weeks
  Change in fat mass, as measured using dual-energy x-ray absorptiometry, from baseline to after the 12-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Tregellas, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States